CLINICAL TRIAL: NCT01241994
Title: Automatic Adaptive System Dialysis (AASD) for Dialysis Related Hypotension and Intolerance: a Prospective Long-term Multicenter Study
Brief Title: Automatic Adaptive System Dialysis (AASD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Other Study IDs: 106/2004/U/Oss
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Dialysis Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- basal hemodialysis (No Intervention)
- AASD (Active Comparator)
  Interventions: Other: AASD dialysis technique

INTERVENTIONS:
Other: AASD dialysis technique
  Arms: AASD

SUMMARY:
AASD is a new dialysis technique based on the use of a mathematical model of intradialytic solutes and fluid kinetic, for the automatic elaboration of dialysate sodium and ultrafiltration rate profile. The aim of dialysate sodium and ultrafiltration rate profile is to obtain the higher stabilization of intradialytic extra cellular compartment, in consideration of end session targets: body weight and final patient's natremia. In this multicenter prospective controlled randomized trial the primary end-point is the clinical efficiency validation of AASD on intradialytic hypotension but also on thirst, cramps, headache, nausea, vomiting, hypotensive events observed in basal treatment (HD or HDF).

ELIGIBILITY:
Inclusion Criteria:Patients in HD/HDF (bicarbonate dialysis/hemodiafiltration) for at least 6 months

* aged more than 18 years
* on chronic thrice-weekly HD
* symptomatic hypotension during at least 30% of dialysis sessions on basal treatment in the last month before admission or/and 1 hypotension /week
* disequilibrium symptoms (cramps, headache, nausea, vomiting, hypotensive events) in at least 30% of dialysis sessions on basal treatment
* dialysis session time: 4 hours (as much as possible)
* Signed inform consent form
* Patients having no vascular access related problems (bi-ponction, blood flow rate 300ml/min)

Exclusion Criteria: Patients in a pregnant state

* Patients whose life expectancy is less than study period
* Patients with progressive acute pathology (neoplasia…)
* Patients included in an other protocol
* Psychiatric patients or patients unable to consent or unable to follow the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
number of intradialytic hypotensive events

SECONDARY OUTCOMES:
percentage of dysequilibrium symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- policlinico S. Orsola, Bologna, Italy

REFERENCES:
- [Result] Coli L, Ursino M, Dalmastri V, Volpe F, La Manna G, Avanzolini G, Stefoni S, Bonomini V. A simple mathematical model applied to selection of the sodium profile during profiled haemodialysis. Nephrol Dial Transplant. 1998 Feb;13(2):404-16. PMID 9509454
- [Result] Ursino M, Coli L, Brighenti C, De Pascalis A, Chiari L, Dalmastri V, La Manna G, Mosconi G, Avanzolini G, Stefoni S. Mathematical modeling of solute kinetics and body fluid changes during profiled hemodialysis. Int J Artif Organs. 1999 Feb;22(2):94-107. PMID 10212044